CLINICAL TRIAL: NCT01730365
Title: Discrimination of Benign and Malignant Human Tissue During Percutaneous Interventions Using Optical Spectroscopy Techniques
Brief Title: Optical Detection of Malignancy During Percutaneous Interventions
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: NL40578.031.12
Record Dates: First submitted 2012-10-04; First posted 2012-11-21 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Coin Lesion; Colon Cancer Liver Metastasis; Breast Cancer
Keywords: spectroscopy; tumour; biopsy; malignancy
MeSH Terms: conditions — Solitary Pulmonary Nodule; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biopsies are taken from the enrolled patients and these biopsies are send to the pathology department for histopathological analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Histological biopsy procedures: Patients with a suspicious lesion in lung or liver or breast who are planned for a standard core biopsy procedure. And patients planned for percutaneous RFA (Radiofrequency Ablation) of colorectal liver metastasis
  Interventions: Procedure: Core biopsy procedure

INTERVENTIONS:
Procedure: Core biopsy procedure — Core biopsy of suspicious lesion in lung, liver, breast, or colorectal liver metastasis.
  Other Names: Histological biopsy procedure; Standard biopsy procedure

SUMMARY:
Investigation of application possibilities of optical spectroscopy within the field of oncology. Optical spectroscopy enables the possibility to specifically differentiate between different (human) tissues. The hypothesis is that incorporation of this technique into existing medical devices (e.g. biopsy needle) would enlarge the accuracy and reliability of these devices. The purpose is to improve and speed up the diagnostics and therapy of the malignancies.

DETAILED DESCRIPTION:
Primary Objective:

In this observational study the investigators aim to evaluate whether optical spectroscopy can correctly diagnose malignant tissue in the existing clinical workflow of percutaneous interventions in lung, liver, and breast.

Secondary Objective:

During the measurement procedure, possible improvements of the measurement hardware will be recorded. Analysis of this documentation will provide information for possible alterations of hardware design for improved clinical applicability in the future. Special attention will be paid to observe how the procedure fits in the standard workflow of the radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspicious lesion in lung or liver who are scheduled for a standard core biopsy procedure
* Patient planned for percutaneous RFA of colorectal liver metastasis
* Written informed consent
* Patients ≥ 18 years old
* Breast patients with a BIRADS score 4 or 5

General Exclusion criteria:

* Patients who have higher risk of bleeding
* Patients with suspected sensitivity to light; e.g. patients who have had photodynamic therapy

Breast Specific Exclusion criteria:

* Patients who have a history of breast cancer and/or who have received prior chemotherapy, endocrine therapy, or radiation therapy
* Patients who have breast implants
* Patients needing a stereotactic breast biopsy (i.e. non palpable-, ultrasound opaque lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are all patients, who are scheduled for a standard core biopsy of lung, liver or breast; or percutaneous RFA of liver in the Netherlands Cancer Institute (NKI-AvL), Amsterdam, The Netherlands. In the enrollment process the "patient informatie" will be used and the informed consent must be signed prior to the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Differentiation between normal and malignant tissue | Day 0
  Statistical analysis of the difference between diffuse reflectance spectra obtained at normal and malignant measurement locations

CONTACTS AND LOCATIONS:
Overall Officials: Theo Ruers, MD, Principal Investigator — Nederlands Kanker Instituut/Antonie van leeuwenhoek Ziekenhuis
Locations (1):
- Nederlands Kanker Instituut/Antonie van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] de Boer LL, Bydlon TM, van Duijnhoven F, Vranken Peeters MTFD, Loo CE, Winter-Warnars GAO, Sanders J, Sterenborg HJCM, Hendriks BHW, Ruers TJM. Towards the use of diffuse reflectance spectroscopy for real-time in vivo detection of breast cancer during surgery. J Transl Med. 2018 Dec 19;16(1):367. doi: 10.1186/s12967-018-1747-5. PMID 30567584